CLINICAL TRIAL: NCT04292340
Title: The Efficacy and Safety of Anti-SARS-CoV-2 Inactivated Convalescent Plasma in the Treatment of Novel Coronavirus Pneumonia Patient (COVID-19) : An Observational Study
Brief Title: Anti-SARS-CoV-2 Inactivated Convalescent Plasma in the Treatment of COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Responsible Party: Principal Investigator, Hongzhou Lu, professor, Shanghai Public Health Clinical Center
Other Study IDs: Anti-SARS-CoV-2
Record Dates: First submitted 2020-02-25; First posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Coronavirus
Keywords: Plasma transfusion; Coronavirus
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is still no effective antiviral drugs and vaccines against SARS-CoV-2 yet now. This is an obsevational study, the investigators collected the clinical information and clinical outcomes of the COVID-19 patients using anti-2019-nCoV inactivated convalescent plasma.The study is to evaluate the efficacy and safety of anti-2019-nCoV inactivated convalescent plasma in the treatment of COVID-19 pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* The participants were diagnosed as COVID-19;
* Participants received anti-SARS-CoV-2 inactivated convalescent plasma
* Written the informed consent.

Exclusion Criteria:

* Participants lacked detailed medical history

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants received anti-SARS-CoV-2 inactivated convalescent plasma
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The virological clearance rate of throat swabs, sputum, or lower respiratory tract secretions at day 1 | 1 day after receiving plasma transmission
  The SARS-CoV-2 nuclei acid was quantified using RT-PCR
The virological clearance rate of throat swabs, sputum, or lower respiratory tract secretions at day 3 | 3 days after receiving plasma transmission
The virological clearance rate of throat swabs, sputum, or lower respiratory tract secretions at day 7 | 7 days after receiving plasma transmission
Numbers of participants with different Clinical outcomes | From receiving plasma transmission to 4 weeks
  Clinical outcomes include death, critical illness, recovery

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 4 weeks after receiving plasma transmission

CONTACTS AND LOCATIONS:
Overall Officials: Hongzhou Lu, Ph.D, Principal Investigator — Shanghai Public Health Clinical Center
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China